CLINICAL TRIAL: NCT00342433
Title: Intraprostatic Androgenicity in Relation to Circulating Levels of Hormones and Polymorphisms of Hormone-Related Genes: A Methodologic Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999025; OH99-C-N025
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Prostate
Keywords: Androgens; Serum; Tissue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Localized Prostate Cancer cases: Cases enrolled between Jan 2000 and Apr 2004 at five locations. Study subject eligibility: Age >=18; scheduled for radical prostatectomy; and newly diagnosed with localized prostate cancer.

SUMMARY:
Although compelling evidence from laboratory studies suggests that androgens play a major role in prostate carcinogenesis, epidemiologic studies in humans (almost exclusively serologic studies) have been unable to confirm the hormonal hypothesis. The major limitation in these serologic studies may stem from difficulty in measuring androgenicity directly at the target site - the prostate. If circulating hormones do not reflect intraprostatic hormone levels or androgenicity, it is not clear how we should interpret results from serum/plasma measurements, and it is unlikely that future serologic studies can clarify the role of hormones in prostate cancer etiology.

This study is a comprehensive methodologic study designed to collect venous blood and prostatic tissue from 650 patients (100 Chinese, 500 American, and 50 Italian) undergoing prostatic surgery (radical prostatectomy, cystoprostatectomy, or transurethral resection of the prostate) in order to correlate prostate tissue with serum hormone levels, and with polymorphisms of hormone-related genes (including the androgen receptor and SRD5A2, the gene encoding 5-alpha-reductase Type II), and to examine characteristics (such as age, smoking, body size) that might affect serum-tissue correlation. We plan to study the following hormones: testosterone, dihydrotestosterone, androstenedione, androstandediol glucuronide, estradiol, estrone, and estrone sulfate. Levels of androgen receptor and its associated protein in prostatic tissue will also be measured to provide a better estimate of total intraprostatic androgenicity. We also plan to collect saliva from 100 of these cases in the Washington, D.C. area and 100 of these cases in China, to assess whether this non-invasive tissue collection method is valid for hormone measurements. Finally, urine collection from 100 of these Chinese men is planned for study of androgen metabolites.

Additionally, we plan to include 200 Chinese subjects for blood collection without tumor tissue for gene polymorphism studies, bringing the total number of subjects enrolled to 850.

For the 650 subjects providing prostate tissue, 30-ml of fasting blood will be collected for hormone and polymorphism analyses, and tissue will be collected at surgery. A 15-minute interview will be conducted to elicit information on demographic characeristics, tobacco and alcohol use, body size, and medical history.

The proposed methodologic study will be the first of its kind to investigate androgenicity in target tissues directly, and the correlation of target tissue androgenicity with circulating levels of hormones and polymorphisms of hormone-related genes in a well-designed epidemiologic study. This study will provide critical information to guide future analytic studies on hormones and prostate cancer.

DETAILED DESCRIPTION:
Although androgens (male hormones) have been the central hypothesis in prostate cancer etiology for decades, epidemiologic studies in humans have not been able to confirm this hormonal hypothesis. Most of the studies used sere (blood) to examine the relationships of circulating hormones with subsequent prostate cancer risk. However, it is possible that circulating levels of hormones may not reflect intraprostatic and androgenic activity accurately.

To gain further insights and to provide directions for future epidemiologic studies, the National Cancer Institute (NCI) is conducting a comprehensive methodological study called Intraprostatic androgenicity in relation to circulating levels of hormone and polymorphisms of hormone-related genes: a methodologic study. The specific aims of this study are:

* to correlate circulating levels of androgens and estrogens with tissue levels (including testosterone, DHT, DHT sulfate, androstenedione, androstanediol glucuronide, estradiol, estrone, and estrone sulfate);
* to determine whether the serum-tissue correlation is mediated by age, race, and selected epidemiologic factors, such as smoking and body size;
* to determine whether tissue hormone levels correlate with polymorphisms of certain hormone-related genes, including androgen receptor (AR) and SRD5A2; and
* to correlate circulating levels of hormones with intraprostatic androgenicity, as defined by the combined levels of tissue hormones, androgen receptor, and its associated protein (ARA70).

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must be over age 18.

Subjects must have a newly diagnosed prostate disease or condition.

Subjects must not currently take hormones.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer cases diagnosed at the collaborating centers
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 1999-05-05 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Intraprostatic hormone concentrations | Cross-sectional
  comparisons between circulating and intraprostatic hormones

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Cook, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - GW University Medical Center GW Hospital Center, Washington D.C., District of Columbia
  - Doctors Community Hospital, Lanham, Maryland
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fairfax Hospital, Falls Church, Virginia
- Shanghai Cancer Institute, Shanghai, China

REFERENCES:
- [Background] Hsing AW. Hormones and prostate cancer: where do we go from here? J Natl Cancer Inst. 1996 Aug 21;88(16):1093-5. doi: 10.1093/jnci/88.16.1093. No abstract available. PMID 8757182
- [Background] Montie JE, Pienta KJ. Review of the role of androgenic hormones in the epidemiology of benign prostatic hyperplasia and prostate cancer. Urology. 1994 Jun;43(6):892-9. doi: 10.1016/0090-4295(94)90163-5. PMID 7515207
- [Background] Vatten LJ, Ursin G, Ross RK, Stanczyk FZ, Lobo RA, Harvei S, Jellum E. Androgens in serum and the risk of prostate cancer: a nested case-control study from the Janus serum bank in Norway. Cancer Epidemiol Biomarkers Prev. 1997 Nov;6(11):967-9. PMID 9367072